CLINICAL TRIAL: NCT05608304
Title: The Effectiveness and Acceptability of Formal Versus Informal Mindfulness Among University Students With and Without Recent Nonsuicidal Self-injury: An Online, Parallel-group, Randomized Controlled Trial
Brief Title: Formal Versus Informal Mindfulness Among University Students With and Without Recent Nonsuicidal Self-injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Social Sciences and Humanities Research Council of Canada (Other)
Responsible Party: Principal Investigator, Nancy Heath, Distinguished James McGill Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 435-2022-0426
Record Dates: First submitted 2022-10-06; First posted 2022-11-08 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Nonsuicidal Self-injury; Mindfulness; Stress; Well-Being
Keywords: Nonsuicidal Self-injury; Mindfulness; Stress; Well-Being; University Students
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Formal mindfulness induction (Experimental)
  Interventions: Behavioral: Formal mindfulness induction
- Informal mindfulness induction (Experimental)
  Interventions: Behavioral: Informal mindfulness induction
- Active control task (Active Comparator)
  Interventions: Behavioral: Active control task

INTERVENTIONS:
Behavioral: Formal mindfulness induction — The formal mindfulness induction will consist of a 10-minute audio recording of a sitting meditation, guiding the participant to consciously and repeatedly bring their attention to their breath and inner experience with nonjudgmental acceptance.
  Arms: Formal mindfulness induction
Behavioral: Informal mindfulness induction — The informal mindfulness induction will consist of on-screen instructions guiding participants through the completion of four routine tasks (washing hands, drinking water, laying down, listening to music) with mindful awareness and acceptance over the course of 10 minutes.
  Arms: Informal mindfulness induction
Behavioral: Active control task — Participants assigned to the active control condition will be prompted to download a single-page document containing 100 letters, numbers, and symbols, and a grid of 100 boxes. Following along with a guided audio, participants will be instructed to place all of the characters in the grid in a specific order over the course of 10 minutes. A version of this task has been used in previous studies by our team (Carsley & Heath, 2019; Petrovic et al., 2022) and has been shown not to impact mindfulness levels, and was thus deemed an appropriate neutral attention task for this study.
  Arms: Active control task

SUMMARY:
The present study will use a randomized controlled design to investigate group differences between students with and without a history of nonsuicidal self-injury (NSSI) in response to a single-session mindfulness induction across conditions (formal mindfulness induction, informal mindfulness induction, active control task) in terms of the intervention's acceptability and effectiveness. Effectiveness will be inferred via pre-post changes in state mindfulness, state stress, and state well-being.

DETAILED DESCRIPTION:
As university students have reported increasing levels of stress and difficulty coping with the challenges of university, student services have had to consider alternative approaches to meet the demand for student support. Thus, universities have moved beyond traditional mental health services to instructional, resilience-building approaches to enhance students' resilience and coping capacity. Mindfulness is a common foundation of these approaches due to the substantial evidence demonstrating the mental health and well-being benefits of mindfulness in university students. However, subgroups within the university student population may respond differently to standard mindfulness instruction.

Specifically, research suggests that university students who engage in non-suicidal self-injury (NSSI; the deliberate destruction of one's bodily tissue in the absence of lethal intent) may respond to mindfulness practice differently than students without such a history. Students with a history of NSSI are particularly prone to experiencing challenges in terms of stress, coping, and well-being in the university context. Thus, these students stand to benefit greatly from mindfulness-based programming that is adapted to their needs.

Standard mindfulness instruction generally consists of a combination of formal and informal practice. Formal practices can be conceptualized as structured, sustained attentional guided activities in which mindfulness is practiced within an allotted period of time (e.g., sitting meditation, body scan), whereas informal practices are brief and unstructured, and focus on the experience of one's senses during routine activities (e.g., becoming aware of the feeling of water on one's hands while washing them). Formal practice often requires sustained attention on one's inner experience (i.e., thoughts and emotions) and bodily sensations. Thus, existing difficulties with emotion regulation, self-criticism, and a potentially complex relationship with their body may render this common component of formal mindfulness practice sub-optimally effective among students with a history of NSSI.

By contrast, informal mindfulness strategies that are brief and unstructured may be more appropriate for these students. Nevertheless, only a few studies have attempted to parse out the benefits of formal and/or informal practice, and the results suggest benefits of informal mindfulness that are distinct from formal mindfulness. Furthermore, a recent systematic review examining the benefits of informal mindfulness concluded that informal practices may be more acceptable among those already experiencing difficulties with emotion regulation (e.g., those with recent NSSI engagement). The need for additional studies exploring the potentially differential acceptability and effectiveness of formal and informal mindfulness instruction among groups with unique intrapersonal needs was underscored.

Thus, the present study will use an online, parallel-group, randomized controlled design to investigate group differences between students with and without a history of NSSI in response to a single-session mindfulness induction across conditions (formal mindfulness induction, informal mindfulness induction, active control task) in terms of the intervention's acceptability and effectiveness. Effectiveness will be inferred via pre-post changes in state mindfulness, state stress, and state well-being.

Primary (state mindfulness) and secondary (state stress, state well-being, and acceptability) outcomes will be assessed immediately pre- and post-intervention. It is hypothesized that university students with a history of NSSI will report greater improvements in state mindfulness, state stress, and state well-being (Hypothesis 1a; superiority) as well as greater acceptability (Hypothesis 2a; superiority) in the IM condition, compared to those in the FM and control conditions. University students with a history of NSSI are also expected to report greater improvements in state mindfulness, state stress, and state well-being (Hypothesis 1b; superiority) as well as greater acceptability (Hypothesis 2b; superiority) in the FM condition, compared to those in control condition. Conversely, university students without a history of NSSI are expected to report noninferior improvements in state mindfulness, state stress, and state well-being (Hypothesis 1c; noninferiority) and noninferior acceptability (Hypothesis 2c; noninferiority) in the IM condition, compared to those in the FM. However, these students are expected to report greater improvements in state mindfulness, state stress, and state well-being (Hypothesis 1d; superiority) as well as greater acceptability (Hypothesis 2d; superiority) in the IM and FM conditions, compared to those in the control condition.

ELIGIBILITY:
Inclusion Criteria:

* Current student at the host institution
* 18-29 years old
* Either a history of engaging in NSSI on at least 5 separate days in the last year or no history of ever having engaged in NSSI

Exclusion Criteria:

- Having a history of NSSI that does not fulfill the recency/frequency requirement

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 254 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Change in state mindfulness (as measured by the VAS) | Pre-post intervention (10-minute interval)
  A Visual Analogue Scale (VAS), an instrument commonly used in induction research (e.g., Hessler-Kaufmann et al., 2020), will also be used to assess the momentary experience of five mindfulness facets, as generally described by Baer et al. (2006). Specifically, there will be five researcher-developed VAS items (one for each facet of mindfulness), modelled on the items in the Five Facets of Mindfulness Questionnaire (FFMQ; Baer et al., 2006). Each VAS will consist of a small, unmarked ruler with anchors labeled as "0 = Not true at all" and "10 = Completely true." Instructions will read: "Please indicate the extent to which each statement below accurately reflects your experience in this moment on the corresponding ruler below by dragging the slider," for each of the five facets of mindfulness. Each scale will yield a single subjective state mindfulness facet score from 0 to 10, where a higher VAS score indicates greater state mindfulness (on that facet).

SECONDARY OUTCOMES:
Change in state mindfulness (as measured by the FFMQ-24) | Pre-post intervention (10-minute interval)
  An adaptation of the 24-item Five Facets of Mindfulness Questionnaire (FFMQ-24; Baer et al., 2006; Medvedev et al., 2018) will also be used to measure state mindfulness. Similar to the original FFMQ-24, this questionnaire will consist of five subscales each assessing a specific facet of state mindfulness (observing, describing, acting with awareness, non-judgmental acceptance, and non-reactivity), although items will be adapted to represent experiences in the present moment (rather than more generally). Respondents will be asked to rate each item on a 5-point Likert scale (1 = Not true at all to 5 = Very true). Items will include, "I am 'running on automatic' without much awareness of what I'm doing," and, "I could easily find the words to describe my feelings." Higher scores on each of the adapted FFMQ-24 subscales indicate greater levels of that specific facet of state mindfulness.
Change in state stress (as measured by the VAS) | Pre-post intervention (10-minute interval)
  A VAS for stress (Lesage et al., 2012) will be used to assess state stress. This VAS will consist of a small, unmarked ruler with anchors labeled as "0 = Not stressed at all" and "10 = As bad as it could be." Participants will be asked to "Indicate how stressed you feel in this moment on the ruler below by dragging the slider." The scale yields a single subjective stress score from 0 to 10, where a higher VAS score indicates greater state stress.
Change in state stress (as measured by the PSM-9) | Pre-post intervention (10-minute interval)
  The 9-item Psychological Stress Measure (PSM-9; Lemyre & Tessier, 2003) will also be used to assess state stress. The PSM-9 consists of items such as, "I feel calm," "I feel rushed; I do not seem to have enough time," and, "I feel stressed," rated on an 8-point Likert scale ranging from Not at all (1) to Extremely (8). For the purposes of this study, "in this moment" will be indicated as the timeframe of interest in order to ensure that participants are reporting their state of stress in-the-moment. A higher sum score on the PSM-9 indicates greater state stress.
Change in well-being (as measured by the VAS) | Pre-post intervention (10-minute interval)
  Similar to above, six VAS scales will be used to assess six aspects of state well-being (i.e., whether participants are feeling calm, good, focused, self-critical, distracted, frustrated). Participants will be asked to "Indicate how [calm/good/focused/self-critical/distracted/frustrated] you feel in this moment on the ruler below by dragging the slider" on four separate VAS scales. Each scale yields a single subjective score from 0 to 10, where a higher VAS score indicates greater state well-being (on that specific aspect).
Acceptability (as measured by the TFA questionnaire) | Post-intervention only (5 minutes)
  The Theoretical Framework of Acceptability (TFA) Questionnaire will be used to assess intervention acceptability (Sekhon et al., 2022). This measure assesses the seven components of the TFA (affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, and self-efficacy) which can help identify characteristics of interventions that may be improved (Sekhon et al., 2017). The TFA Questionnaire is adaptable and can be used to evaluate various healthcare interventions. It consists of seven items, each pertaining to one of the components listed above, as well as an eight item that assesses general acceptability. For this trial, the item pertaining to opportunity costs will be omitted as it was deemed not applicable. In its place, an eighth item was created and added to this measure, reflecting concerns around the participant's assigned intervention. All items are rated on 5-point scales; a higher mean score indicates greater acceptability.
Acceptability (as measured by the IMI) | Post-intervention only (5 minutes)
  Subscales of the Intrinsic Motivation Inventory (IMI; Ryan, 1982) will also be used to assess acceptability from a SDT-perspective, as the IMI is intended to assess participants' subjective experience of a target activity in experimental research. For the purposes of this study, four subscales of this measure will be included: interest/enjoyment (5 items; e.g., "I enjoyed doing this activity very much"), perceived competence (5 items; e.g., "I am satisfied with my performance on this activity"), perceived autonomy (6 items; e.g., "I believe I had some choice in how I went about doing this activity"), and value/usefulness (7 items; e.g., "I believe this activity could be of some value to me"). All items are rated on a 7-point Likert scale ranging from Not at all true (1) to Very true (7).

CONTACTS AND LOCATIONS:
Overall Officials: Nancy L. Heath, Ph.D., Principal Investigator — McGill University
Locations (1):
- McGill University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP
URL: https://doi.org/10.1016/j.cct.2023.107109